CLINICAL TRIAL: NCT07177768
Title: Acute Effects of Prolonged Walking on Pain, Balance and Posture in Individuals With Hallux Valgus Deformity
Brief Title: Acute Effects of Prolonged Walking on Hallux Valgus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Kübra Alpay, Lecturer of Pysiotherapy and Rehabilitation Department, Bezmialem Vakif University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KA25-2
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hallux Valgus Group (Experimental): Individuals with hallux valgus deformity
  Interventions: Other: Prolonged walking
- Control Group (Other): Healthy controls
  Interventions: Other: Prolonged walking

INTERVENTIONS:
Other: Prolonged walking — walking on a treadmill for 60 minutes

SUMMARY:
Hallux valgus is a progressive foot deformity characterized by lateral deviation of the great toe and medial displacement of the first metatarsal head. While pain is a common symptom among individuals with HV, alterations in plantar pressure distribution and impaired balance are also frequently observed. These symptoms and biomechanical changes can negatively impact posture and gait mechanics. The aim of this study is to investigate the acute effects of prolonged walking on pain, balance, posture, and gait in individuals with hallux valgus deformity.

DETAILED DESCRIPTION:
Hallux valgus is a progressive foot deformity commonly seen in adults. Patients typically report pain, most prominently in the first metatarsophalangeal joint, which is often exacerbated by weight-bearing activities such as walking. Due to the deformity, alterations in plantar pressure distribution occur, which in turn affect plantar sensory input and postural control. This may lead to decreased postural stability, impaired balance, and compromised control during walking. HV is also thought to accelerate biomechanical changes that negatively impact gait patterns. The aim of this study is to evaluate the acute effects of prolonged walking on pain, balance, posture, and gait in individuals with hallux valgus deformity. A total of 32 participants, including individuals with HV and healthy controls, will be included in the study. All participants will walk on a treadmill for 60 minutes. Assessments will be conducted at three time points: before walking, immediately after walking, and 20 minutes post-walking.

ELIGIBILITY:
Inclusion Criteria:

Hallux Valgus Group Criteria:

* Individuals aged between 18 and 55 years
* Being diagnosed with hallux valgus

Control Group Criteria:

* Individuals aged between 18 and 55 years
* Classified as grade A according to the Manchester Scale
* Being a volunteer

Exclusion Criteria:

* History of previous foot or ankle surgery
* Having a systemic diseases
* Having a neurological disorders
* Having a vestibular pathologies that may affect balance

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline, immediately after intervention, 20 minutes after intervention
  Pain intensity will be evaluated with visual analog scale (VAS). Patients will be asked to mark the intensity of the pain they feel on a 10 cm line, where "0" means no pain and "10" means the worst pain.
Pressure pain threshold | Baseline, immediately after intervention, 20 minutes after intervention
  It will be measured with algometer. Higher values indicate a higher perceived pain threshold.
Single-leg stance test | Baseline, immediately after intervention, 20 minutes after intervention
  The single leg stability will be assessed by using Biodex Balance System® (Biodex Medical Systems, Inc. USA). Low values of the stability index indicate better balance and stability.
Postural Assessment | Baseline, immediately after intervention, 20 minutes after intervention
  Posture will be assessed using mobile application. It marks and measures angles at the ear, shoulder, anterior superior iliac spine (ASIS), knee, and ankle alignment to identify any pathological deviations or asymmetries.
Gait analysis | Baseline, immediately after intervention, 20 minutes after intervention
  Gait analysis will be performed using mobile application. Subjects are asked to walk at their normal walking speed over a 10-meter surface, and measurements are taken using video recording and evaluated using the software. The assessment records right and left step lengths, double step length, stride width, and walking speed.

CONTACTS AND LOCATIONS:
Overall Officials: Ozgur Serbest, Pt, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Eyup, Turkey (Türkiye)